CLINICAL TRIAL: NCT05578404
Title: The Effect of High Oral Loading Dose of Cholecalciferol in Non-Alcoholic Fatty Liver Disease Patients
Brief Title: High Oral Loading Dose of Cholecalciferol in Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2022
Record Dates: First submitted 2022-10-08; First posted 2022-10-13 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): 50 patients will receive the standard conventional therapy in addition to a placebo for 4 months.
  Interventions: Drug: Placebo
- Vit D Group (Active Comparator): 50 patients were given the standard conventional therapy plus cholecalciferol. Cholecalciferol was given as a high oral loading dose of 300,000 IU followed by a daily oral dose of 800 IU for 4 months.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Vit D is a fat-soluble vitamin, provided by sunlight and activated by kidneys and liver.
  Arms: Vit D Group
Drug: Placebo — matching placebo to Vit D
  Arms: Control Group

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a metabolic disorder with high prevalence in patients suffering from chronic liver diseases [1]. NAFLD is characterized by the accumulation of > 5% of fat deposits in hepatocytes (hepatic steatosis) with no known other reasons for steatosis as excessive alcohol intake.The global prevalence of NAFLD differs depending on the population reaching 13% in Africa, 32% in the Middle East, and 30 % in the United States

ELIGIBILITY:
Inclusion Criteria:

* Either male or female adult patients (>19 years) with fatty liver diagnosis by using upper abdominal ultrasound echography (US) and with type II diabetes diagnosed according to American Diabetes Association (ADA) 2019 criteria and treated with metformin

Exclusion Criteria:

* pregnant and/or lactating women, excessive alcohol use (defined as an average alcohol intake of> 30 g per day in men and > 20 g per day in women),
* Other etiology of chronic liver diseases such as viral hepatitis, drug-induced hepatitis, autoimmune hepatitis, patients suffering from chronic kidney disease, and hyper/hypoparathyroidism.
* Hypersensitivity to cholecalciferol, hypercalcemia, patients taking supplementation with vitamin D, and calcium.
* Medications affecting calcium/vitamin D metabolism (as anticonvulsants, glucocorticoids, and antacids).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose (FBG mg/dl) | 4 months
Glycated hemoglobin (HbA1C%) | 4 months
Fasting insulin (mU/L). | 4 months
Alanine transaminase (ALT U/L) | 4 months
Aspartate transaminase (AST U/L) | 4 months
Albumin (g/dl) | 4 months
Gamma-glutamyl transferase (GGT U/L) | 4 months
Alkaline phosphatase (ALP U/L) | 4 months
Lipid profile: Low-density lipoprotein (LDL-C mg/dl), High-density lipoprotein (HDL-C mg/dl) | 4 months
Lipid profile: Triglycerides (TG mg/dl) | 4 months
Lipid profile: Total cholesterol (TC mg/dl) | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt